CLINICAL TRIAL: NCT07268209
Title: Validation of a Score for Supplementation Needs of Vitamins, Micronutrients and Proteins After Bariatric Surgery
Acronym: BARSCORE
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Universitari de Bellvitge - IDIBELL (Unknown)
Responsible Party: Principal Investigator, Javier Osorio, Head of Esophago-gastric and Bariatric Surgery Unit, Hospital Universitari de Bellvitge
Other Study IDs: HUB-CIR-BARSCORE
Record Dates: First submitted 2025-09-13; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Obesity &Amp; Overweight; Bariatric Surgery; Bariatric Surgery Complication
Keywords: Bariatric surgery; Nutritional supplementation; Vitamin deficiency; Clinical score validation
MeSH Terms: conditions — Obesity; Overweight; Avitaminosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ABSTRACT Obesity is, nowadays, a pandemic. The treatment of patients affected by obesity is very complex and requires the synergy of a multidisciplinary team that addresses the problem in its different spheres. Among the available treatment options, surgery remains the most effective in the long term. Among surgical techniques, there are different types based on different mechanisms. Among them, hypoabsorptive techniques, which are the most effective, can lead to malnutrition and vitamin deficiencies, so the creation of a standardized score -similar to Clavien-Dindo- could be a simple, reproducible tool with sufficient clinical relevance to allow comparison of nutritional outcomes between different surgical techniques.

Hypothesis: The BARSCORE score will allow estimation of supplementation needs for vitamins, micronutrients and proteins after bariatric surgery.

Objectives: To validate a score in bariatric surgery that grades supplementation needs by relating them to patient characteristics and the proposed surgical technique.

Methodology: observational, longitudinal, multicenter study. The study sample will consist of patients who underwent bariatric surgery between January 2015 and December 2021 in participating centers (Appendix 1).

Patients will be divided into three groups based on the surgery performed and the score will be applied. Subsequently, surveys will be conducted to evaluate the score and cases for applying the score.

For statistical analysis, Spearman's correlation test will be used to verify the consistency of the score and a two-way ANOVA analysis to measure its concordance.

DETAILED DESCRIPTION:
INTRODUCTION Morbid obesity is considered the great epidemic of this century. It is the leading cause of non-traumatic death in the Western population and is progressively affecting developing countries. In the latest epidemiological studies, it is estimated that in Spain more than 15% of the population is overweight, and approximately 5% suffer from morbid obesity.

The treatment of morbid obesity is multidisciplinary, ranging from changes in lifestyle habits and diet to surgery. Among all available therapeutic options, bariatric surgery is the only cost-effective long-term treatment for patients with morbid obesity. It offers better results than pharmacological treatments and lifestyle changes. Furthermore, it has been shown to reduce and improve comorbidities, improve quality of life, reduce the risk of cardiovascular diseases and mortality, and improve quality of life.

There are currently several standardized bariatric surgical techniques. These techniques can be restrictive such as vertical gastrectomy (VG), hypoabsorptive such as duodenal switch (DS) and single-anastomosis duodeno-ileal bypass with sleeve gastrectomy (SADI-S), or mixed such as gastric bypass (GBP). Their indication will depend on factors such as the patient's BMI, metabolic comorbidities, or the surgical team's experience, among others. All of them have proven to be safe in experienced teams, with mortality rates equal to or less than 0.5% and morbidity less than 10%.

Although postoperative risks are low, they must be considered along with the potential benefits of surgery on an individual basis and as accurately as possible in each case. This allows the decision to perform surgery to be made consensually with the patient based on objective data.

One of the main risks, especially of mixed and hypoabsorptive techniques, is the risk of malnutrition and vitamin deficiencies. This complication is recorded in the literature in a heterogeneous and non-comparable manner. Articles documenting levels of nutrients, vitamins, and trace elements in blood during follow-up after bariatric surgery are complex to assess since data collection is not performed in a standardized way and it is not specified whether blood levels are with or without supplementation or the supplementation dose received; making them non-uniform and difficult to compare with each other.

A classification based on the therapeutic effort needed to resolve nutritional deficits (similar to the concept of the Clavien-Dindo classification for short-term post-surgical complications) could have the advantage of simplicity, reproducibility, and sufficient clinical relevance to allow comparison between different surgical techniques. This score could be evaluated along with efficacy (amount of weight lost and resolution of comorbidities) and morbidity (short and long-term complications) to assess the pros and cons of each surgical technique for each patient profile.

The bariatric surgery, endocrinology, and nutrition teams from HUB, HCP, and VHG hospitals reached consensus on a score for predicting therapeutic effort in supplementation after bariatric surgery. The objective of the present study is to retrospectively validate its utility and reproducibility in patients operated on for vertical gastrectomy, gastric bypass, duodenal switch, and single-anastomosis duodenal switch with a minimum of two years of clinical and analytical follow-up.

HYPOTHESIS The BARSCORE score will allow estimation of supplementation needs for vitamins, micronutrients, and proteins after bariatric surgery.

The BARSCORE score will be a coherent score, so that more complex surgeries will have higher scores in the score with a Spearman correlation test with p <0.05.

The BARSCORE score will be a score with a high level of concordance since different investigators from each center will score the presented cases in the same way, obtaining a two-way analysis of variance with p <0.05.

The BARSCORE score will be an easy-to-apply score since it will obtain a percentage of favorable results greater than 70% in the score evaluation survey.

GENERAL OBJECTIVE To validate a score in bariatric surgery that grades supplementation needs by relating them to patient characteristics and the proposed surgical technique.

SPECIFIC OBJECTIVES

Demonstrate the coherence of the score after comparing different types of surgical techniques with different complexity and their obtained score.

Verify concordance through responses obtained by investigators from each center in the case survey to apply the score.

Verify ease of application through the percentage of favorable responses obtained in the score evaluation survey by participating investigators from each center.

METHODS Study Design Observational, multicenter (participating centers in Appendix 1), longitudinal study based on the medical records of a cohort of patients operated on for primary laparoscopic bariatric and metabolic surgery from January 2015 to October 2022, in participating centers.

Procedure:

Patient recruitment: inclusion of patients in the multicenter online database. Division of patients into three groups according to the surgery performed (vertical gastrectomy, gastric bypass, and single and double anastomosis duodenal switch) and categorization of patients using the supplementation needs score.

Determine score coherence: comparison of score results between different groups of surgical techniques based on their complexity using Spearman's correlation coefficient.

Verify score concordance (reproducibility): at least two investigators from each center will answer the case survey to apply the score. Subsequently, a two-way ANOVA analysis will be performed on the case survey after applying a normal distribution transformation of the percentage of correct answers (Appendix 2).

Verify ease of score application with responses from at least two investigators from each center to a survey about the complexity and utility of the score, performing a descriptive analysis of the results.

Study Population

Patients undergoing primary minimally invasive bariatric surgery from the population area of all participating centers, between 18 and 65 years of age, in the period from January 2015 to July 2022.

Inclusion criteria: Patients operated on for primary laparoscopic bariatric surgery using vertical gastrectomy, gastric bypass, duodenal switch, or single-anastomosis duodenal switch (SADI-S) techniques between 2015 and 2022 in participating centers, with minimum 2-year follow-up, with analytical control and evaluation by endocrinologist and dietitian/nutritionist.

Exclusion criteria: Patients operated on for revisional surgery or with less frequent techniques such as single-anastomosis gastric bypass or intestinal bipartition. Patients operated on via open approach or requiring conversion to open approach during surgery. Patients with loss to follow-up.

EXPERIMENTAL TREATMENT:

Primary laparoscopic bariatric or metabolic surgery.

ASSESSMENT CRITERIA:

The study will consist of validating the score through these three criteria:

Number of patients in each score category after laparoscopic bariatric surgery. Using 1-2-3 Degree of score coherence based on observed differences between different techniques.

Degree of concordance (reproducibility) of assigning each patient to their corresponding category among different professionals.

Degree of ease according to the opinion of professionals answering the evaluation survey.

SAMPLE SIZE DETERMINATION:

This is an exploratory study in which the sample size cannot be numerically justified in usual terms. In fact, reliable data on the expected magnitude of differences are currently unknown, given that homogeneous results regarding the risk of malnutrition and vitamin deficiencies are not available in the literature. As a consequence, formal numerical calculation is not possible.

At least 1200 patients will be included, corresponding to patients from the study period, from January 2015 to October 2022, at the main investigational center (Bellvitge Hospital). This number seems reasonable in an exploratory context, supported by additional references with similar sample sizes in this field (for example, Clavien-Dindo). Furthermore, conducting this study is especially relevant, as it may provide important results for the proposed objectives and lay the groundwork for future confirmatory studies.

STATISTICAL CONSIDERATIONS:

Categorical variables will be presented as number of cases and percentages, and continuous variables with mean and standard deviation.

Initial risk factors to be included in the model are composed of sociodemographic data such as age, sex, and individual BMI, comorbidities, type of bariatric surgery, as well as its complications.

For coherence, a Spearman correlation test will be applied, taking a p value <0.05 as significant.

For concordance, a two-way analysis of variance (two-way ANOVA) will be performed assuming assumptions of normality and homoscedasticity, with p values <0.05 considered statistically significant.

For ease of application, a descriptive analysis of the score evaluation survey results will be performed using percentages, and values above 70% favorable responses will be considered an easy-to-apply score.

TIMELINE AND WORK PLAN The study will begin in October 2024. Information collection from medical records in the eCRD by participating centers will begin once the Research Ethics Committee approves this study. This activity is expected to be completed by December 2024.

Database cleaning and statistical analyses require at least 3 months (March 2024).

The final report will be available in publication form within six months of completing statistical analyses.

The expected completion date (final report) is October 2025. ETHICAL ASPECTS An electronic data collection questionnaire will be designed in REDCap for this study. The data collection system will be online, via web, and data will be stored on an IDIBELL server with high security measures. Each investigator from each center will have particular access protected with a password. Their access will allow them to enter and correct data from patients at their center, but not from other centers.

Since this is a study based on information collected from medical records, in an anonymized manner, and due to the difficulty of contacting patients and the number of patients lost to follow-up, written consent will not be requested.

Patients will be identified by an identification number assigned when entering them into the database, removing the medical record number and date of birth, thus making identity tracing difficult. Only an IDIBELL statistician and a reference person from each center will have access to the correlation between identification number and medical record number, governed by article 14 GDPR and Additional Provision 17 of Organic Law 3/2018 on Personal Data Protection and Guarantee of Digital Rights.

A document with authorization from the clinical research ethics committee is attached.

RESOURCES AND INFRASTRUCTURE The resources and infrastructure of each participating hospital will be used for patient recruitment and treatment, according to usual surgical activity. The computer infrastructure will be provided by IDIBELL through the online database where results from all patients will be collected and analyzed.

PROJECT BENEFITS A score can be created and validated that will allow measuring and quantifying the need for supplementation after bariatric surgery and, similarly, quantify patients' nutritional deficits in a standardized and comparable manner, thus making comparison between techniques, surgeons, and centers possible.

This score will provide a new way to add objective information to assess the pros and cons of each surgical technique applied individually to each patient. So that to assess the pros we will have total weight loss percentage (%TWL) and resolution of comorbidities, and for the cons, short-term surgical complications using Clavien-Dindo and long-term complications using the Barscore score.

All of this will contribute to providing more information to the patient for shared informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on for primary laparoscopic bariatric surgery using vertical gastrectomy, gastric bypass, duodenal switch, or single-anastomosis duodenal switch (SADI-S)
* Techniques between 2015 and 2022 in participating centers.
* Minimum 2-year follow-up.
* Analytical control and evaluation by endocrinologist and dietitian/nutritionist.

Exclusion Criteria:

* Patients operated on for revisional surgery.
* Patients operated with less frequent techniques such as single-anastomosis gastric bypass or intestinal bipartition.
* Patients operated on via open approach or requiring conversion to open approach during surgery.
* Patients with loss to follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary minimally invasive bariatric surgery from the population area of all participating centers, between 18 and 65 years of age, in the period from January 2015 to July 2022.
Sampling Method: Probability Sample
Enrollment: 4514 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09-13 (Actual)

PRIMARY OUTCOMES:
Score coherence | Baseline score measurement at inclusion in the study
  Measure: Spearman correlation coefficient between surgical complexity and BARSCORE score (0: no supplements, I protocol, II oral supplements, III parenteral supplements, IV mild malnutrition, V severe malnutrition). Higher values of the score indicate a greater need for supplementation.
  Success criteria: p <0.05
Score Concordance (reproducibility) | Through study completion, an average of 6 months
  Measure: Two-way ANOVA analysis of responses from different investigators on standardized cases. The investigators will be given a list of cases where they have to apply the BARSCORE score (0: no supplements, I protocol, II oral supplements, III parenteral supplements, IV mild malnutrition, V severe malnutrition).
  Success criteria: p <0.05
Ease of Application | Through study completion, an average of 6 months
  Measure: Percentage of favorable responses in the evaluation survey Success criteria: >70% favorable responses

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Privacy and Ethical Constraints: The protocol explicitly states that patient data will be anonymized and stored on secure IDIBELL servers with restricted access. Only specific personnel (IDIBELL statistician and one reference person per center) will have access to patient identifiers.
  Data Governance Structure: Each investigator only has access to their own center's data, not other centers' data, indicating a restrictive data sharing model.

REFERENCES:
- [Background] Collins GS, Reitsma JB, Altman DG, Moons KG. Transparent Reporting of a multivariable prediction model for Individual Prognosis or Diagnosis (TRIPOD): the TRIPOD statement. Ann Intern Med. 2015 Jan 6;162(1):55-63. doi: 10.7326/M14-0697. PMID 25560714
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Guilbert L, Joo P, Ortiz C, Sepulveda E, Alabi F, Leon A, Pina T, Zerrweck C. Safety and efficacy of bariatric surgery in Mexico: A detailed analysis of 500 surgeries performed at a high-volume center. Rev Gastroenterol Mex (Engl Ed). 2019 Jul-Sep;84(3):296-302. doi: 10.1016/j.rgmx.2018.05.002. Epub 2018 Jun 20. English, Spanish. PMID 29933896
- [Background] Anderin C, Gustafsson UO, Heijbel N, Thorell A. Weight loss before bariatric surgery and postoperative complications: data from the Scandinavian Obesity Registry (SOReg). Ann Surg. 2015 May;261(5):909-13. doi: 10.1097/SLA.0000000000000839. PMID 25211265
- [Background] Goitein D, Raziel A, Szold A, Sakran N. Assessment of perioperative complications following primary bariatric surgery according to the Clavien-Dindo classification: comparison of sleeve gastrectomy and Roux-Y gastric bypass. Surg Endosc. 2016 Jan;30(1):273-8. doi: 10.1007/s00464-015-4205-y. Epub 2015 Apr 11. PMID 25861906
- [Background] Zhang L, Tan WH, Chang R, Eagon JC. Perioperative risk and complications of revisional bariatric surgery compared to primary Roux-en-Y gastric bypass. Surg Endosc. 2015 Jun;29(6):1316-20. doi: 10.1007/s00464-014-3848-4. Epub 2014 Oct 8. PMID 25294534
- [Background] Grigaites, Alejandro L., et al. Morbimortalidad posoperatoria en cirugía bariátrica laparoscópica: experiencia en 1020 pacientes. Revista argentina de cirugía. 2014;106(2):1-10.
- [Background] Rubio, Miguel A., et al. Documento de consenso sobre cirugía bariátrica. Rev Esp Obes. 2004;4(7).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT07268209/Prot_SAP_000.pdf